CLINICAL TRIAL: NCT00376077
Title: A Randomized Study of IVIG vs. IVIG With High Dose Methylprednisolone in Rapidly Augmenting Platelet Counts in Childhood ITP.
Brief Title: A Randomized Study of IVIG vs. IVIG With High Dose Methylprednisolone in Childhood ITP.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Manuel Carcao, Staff Haematologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000006180
Record Dates: First submitted 2006-09-12; First posted 2006-09-14 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Thrombocytopenia; pediatric; methylprednisolone; intracranial hemorrhage; intravenous immune globulin
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Intracranial Hemorrhages | interventions — Methylprednisolone; Immunoglobulins, Intravenous; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo and IVIG (Active Comparator): The trial site is blinded to the randomization process. Patients are assigned an arm by a research pharmacist. Patients on this arm receive an infusion of placebo (0.9% NaCl) over one hour. Immediately following this dosing, 1 g/kg IVIG (Gammunex ©) is infused over 2 - 3 hours. Following this treatment, complete blood counts are drawn at:
  * completion of IVIG infusion,
  * 8 hours following the start of the placebo/solumedrol infusion
  * 24 hours following the start of the placebo/solumedrol infusion
  * 72 hours following the start of the placebo/solumedrol infusion
  * 7 days post infusion
  * 21 days post infusion
  Interventions: Drug: Placebo and IVIG
- Methylprednisolone and IVIG (Experimental): The trial site is blinded to the randomization process. Patients are assigned an arm by a research pharmacist.Patients on this arm receive IV Methylprednisolone 30 mg/kg (1 gram maximum) infused over one hour. Immediately following this dosing, 1 g/kg IVIG Gammunex © is infused over 2 - 3 hours. Following this treatment, complete blood counts are drawn at:
  * completion of IVIG infusion,
  * 8 hours following the start of the placebo/solumedrol infusion
  * 24 hours following the start of the placebo/solumedrol infusion
  * 72 hours following the start of the placebo/solumedrol infusion
  * 7 days post infusion
  * 21 days post infusion
  Interventions: Drug: Methylprednisolone and IVIG

INTERVENTIONS:
Drug: Methylprednisolone and IVIG — Combination therapy (IV MP (Solu-Medrol®, Upjohn) 30 mg/kg (max. 1 g) over 1 hour followed by IVIG 1 g/kg (Gamunex Immune Globulin Intravenous [Human], 10%; Bayer)* x 1 dose
  Other Names: Solumedrol
  Arms: Methylprednisolone and IVIG
Drug: Placebo and IVIG — Placebo followed by IVIG 1 g/kg (Gamunex Immune Globulin Intravenous [Human], 10%; Bayer)* x 1 dose
  Arms: Placebo and IVIG

SUMMARY:
Childhood immune thrombocytopenia purpura (ITP) is a disorder characterized by the production of antibodies against platelets, resulting in enhanced destruction of platelets. Most children with ITP present with low platelet counts (PC) but minimal bleeding. Very rarely a child may present with a severe life-threatening bleed, such as a bleed in the head. In this case it is very important that the PC be raised as quickly as possible. The combination of corticosteroids and intravenous gammaglobulin (IVIG) is commonly used in the management of such severe bleeding in children with ITP to quickly raise the PC and yet this treatment combination has not been tested against using IVIG alone. If it is shown that the combination of these agents does result in a quicker rise in PC then when using IVIG alone would support the use of this combination therapy in emergency situations.

As we can not ethically conduct this study in patients with life-threatening bleeds, we plan to study patients with ITP and PC less than 20 X 109/L, but without life threatening bleeding. Eligible patients will be randomized to one of these 2 regimens (IVIG + placebo or IVIG + IV corticosteroids). The study is designed as a double-blind trial, where the patient or the treating physician will not be aware of the regimen that a patient is randomized to. PC's will be measured as a surrogate measure of bleeding risk; bleeding scores (a score generated by observing patients for bleeding symptoms) will be used to grade bleeding severity, and adverse effects to treatment will be monitored by the means of questionnaires throughout the study.

DETAILED DESCRIPTION:
Rarely children with immune thrombocytopenia purpura (ITP) can present with severe or life-threatening bleeding. In these cases it is very important that the platelet count be raised as quickly as possible. Several studies have shown that IVIG and corticosteroids on their own can raise platelet counts, but few studies have examined how the combination of IVIG and corticosteroids compares to IVIG alone in raising platelet counts in childhood ITP. Yet despite the lack of conclusive evidence to indicate that steroids given together with IVIG is more effective, this combination treatment is often given when children present with a life-threatening bleed, e.g. intracranial bleed. In addition to presumed greater effectiveness of giving the two agents together there is also evidence to show that the combination of IVIG with steroids may have other beneficial effects, in addition to greater effectiveness at raising platelet counts. This can include reducing side effects of IVIG.

We propose to compare the effectiveness of the combination of IVIG with corticosteroids to IVIG alone in raising platelet counts in children with ITP and a platelet count less than 20 x 109/L. Patient will be eligible only if they in conjunction with their treating physician have decided to be treated with IVIG. In this way they will require an intravenous regardless of study participation. The primary outcome is the rise in platelet count as reflected by the platelet count at 24 hours.

Hypothesis:

IVMP and IVIG, administered together, will

1. increase the PC faster, and
2. minimize the adverse effects of IVIG, and
3. lead to a more sustained increase in PC (longer time before needing retreatment) If it is shown that the combination of these agents does result in a quicker rise in PC, this would support and justify the use of the combination therapy in emergency situations.

Study Proposal and Methods:

We propose to prospectively evaluate 2 treatment regimens in patients with childhood ITP:

Regimen A: Placebo followed by IVIG 1 g/kg (Gamunex® Immune Globulin Intravenous [Human], 10%; Bayer)* x 1 dose Regimen B: Combination therapy (IV MP (Solu-Medrol®, Upjohn) 30 mg/kg (max. 1 g) over 30 min followed by IVIG 1 g/kg (Gamunex® Immune Globulin Intravenous [Human], 10%; Bayer)* x 1 dose

*Gamunex will be given according to manufacturer's guidelines. Gamunex has been demonstrated to be safely and effectively administered by means of a rapid infusion protocol whereby it can be given over a period of 2 hours (although in some cases it needs to be given at a slower rate over a longer period of time).

ELIGIBILITY:
Inclusion Criteria:

* ages 1-17 yr. followed at participating centers
* diagnosed with primary ITP
* present with a PC < 20 x 10^9/L
* patient and attending physician have decided on treatment of ITP

Exclusion Criteria:

* initial presentation with ITP
* splenectomy
* life-threatening hemorrhage e.g. proven or suspected intracranial hemorrhage (ICH), major gastrointestinal hemorrhage with cardiorespiratory decompensation
* organ-threatening hemorrhage e.g. hemorrhage into the eye
* contraindication to IVIG ( renal disease with creatinine > x 2 upper list of normal )
* contraindication of IV methylprednisolone ( diabetes mellitus, hypertension, peptic ulceration )
* prior failure to attain a PC level over 50 X 109 within 2 weeks of treatment with IVIG of 0.8 to 1 g/kg or IV methyl-prednisolone (max 1 gram ) within 6 months prior to study entry
* co-existing situations that could affect platelet response to therapy e.g. sepsis, fever > 38.5°C ( orally or equivalent), splenomegaly (spleen tip > 2 cm below costal margin), Disseminated Intravascular Coagulation (DIC) - defined by a fibrinogen level < 1.0 g/dL and elevated D-dimer levels, surgery
* pregnancy (a mandatory urine pregnancy test will be obtained on all post-pubescent female patients). Such patients can only be eligible once the urine pregnancy test results are confirmed to be negative.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2005-08; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The rapidity of rise in Platelet Count | The first 24 hours following the administration of therapy

SECONDARY OUTCOMES:
Days to PC falling to < 20 x 109/L | Time frame determined by outcome
Adverse Effects of therapy | 1 week
Quality of life changes over time and between the treatment groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Carcao, MD, Principal Investigator — The Hospital for Sick Children; Victor Blanchette, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Manuscript preparation

REFERENCES:
- [Derived] Carcao M, Silva M, David M, Klaassen RJ, Steele M, Price V, Wakefield C, Kim L, Stephens D, Blanchette VS. IVMP+IVIG raises platelet counts faster than IVIG alone: results of a randomized, blinded trial in childhood ITP. Blood Adv. 2020 Apr 14;4(7):1492-1500. doi: 10.1182/bloodadvances.2019001343. PMID 32282882